CLINICAL TRIAL: NCT06824740
Title: Prevalence of Insufficient Analgesia in Caesarean Section Under Neuroaxial Anesthesia
Brief Title: Prevalence of Insufficient Analgesia in Caesarean Section Under Neuroaxial Anesthesia (PAICAN)
Acronym: PAICAN
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Other Study IDs: PAICAN
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-05

CONDITIONS: Cesarean Section; Analgesia
Keywords: cesarean section; neuraxial anesthesia; pain; analgesia
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pain during caesarean section under neuraxial anesthesia is often underestimated and could be related to perinatal psycholocal disorders.

The implementation of an evidence-based anesthestic management protocol for caesarean sections aims at reducing intraoperative and postoperative pain.

This prospective observational single-center study aims at determining whether this protocol helped to reduce the prevalence of insufficient analgesia in during caesarean sections.

DETAILED DESCRIPTION:
Caesarean surgery is one of the most frequent surgeries around the world and neuroaxial anesthesia is the preferred anesthesia technique in most settings. Still, many women experience pain during caesarean section, and it has implications in their birth experience. The PAICAN study (Prevalence of Insufficient Analgesia in Caesarean Section under Neuroaxial Anesthesia) aims to study how the implementation of a specific protocol of anesthetic management during caesarean section reduces the intraoperative pain and the need of postoperative painkillers.

Other objectives are:

* To study the adherence to the new protocol in our centre
* To understand the mechanisms of the failure of neuraxial anesthesia
* To study the related factors to insufficient analgesia during surgery (demographic, obstetric, anesthetic, etc.).

Hypothesis: the implementation of an anesthestic management protocol for caesarean sections under neuroaxial anesthesia decreases the prevalence of insufficient analgesia during surgery and in the recovery room.

Design: Prospective observational single-center study.

ELIGIBILITY:
Inclusion Criteria:

- Pregnant women aged 18 or more undergoing a caesarean section under neuraxial anesthesia

Exclusion Criteria:

* Non pregnant women
* Women under 18 years old
* General anesthesia as first option for anesthesia
* Refusal to participate in the study
* Women with cognitive impairment or held in an institution by legal or official order

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women undergoing a caesarean section under neuraxial anesthesia in a tertiary hospital in Barcelona (Spain).
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of Insufficient Analgesia during cesarean section | During the cesarean section
  Prevalence of Insufficient Analgesia during cesarean section is a composite variable based on 4 principal variables:
  * Intraoperative Verbal Numeric Scale of Pain (asked intraoperatively)
  * Categorical scale of pain (low, moderate, severe, no pain) (asked intraoperatively)
  * Alternative anesthestic plan (any different anesthetic technique that differs from the initial anesthestic plan)
  * Failure of the initial anesthetic technique (any failure during the whole surgical procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Vilches, MD, Principal Investigator — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided